CLINICAL TRIAL: NCT02886377
Title: The Correlation Between AQP-4 Ab and the Visual Function of Patients With Demyelinating ON at Onset
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiujuan Zhao (Other)
Responsible Party: Sponsor-Investigator, Xiujuan Zhao, doctor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Organization: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Other Study IDs: 2014meky049
Record Dates: First submitted 2016-08-07; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- NMOSD-ON: NMOSD-ON included patients who met the established diagnostic criteria for NMO or NMOSD published by Wingerchuk et al,with AQP4 seropositive according to the results of the AQP4-Ab test.
  Interventions: Biological: blood test of anti-AQP4 antibody
- MS-ON: MS-ON group patients included typical acute demyelinating ON with brain lesions fulfilling the revised McDonald criteria or clinical isolate syndrome (CIS), with AQP4 seronegative according to the results of the AQP4-Ab test.
  Interventions: Biological: blood test of anti-AQP4 antibody
- Healthy controls: Age- and gender- matched healthy controls.
  Interventions: Biological: blood test of anti-AQP4 antibody

INTERVENTIONS:
Biological: blood test of anti-AQP4 antibody — Patients were sub-divided into an AQP4 seropositive group and an AQP4 seronegative group, according to blood test of the AQP4-Ab.

SUMMARY:
To evaluate the optical coherence tomography (OCT), visual field (VF), Visual evoked po-tential(VEP) characteristics between neuromyelitis optica- related optic neuritis (NMOSD-ON) and multiple sclerosis- related ON (MS-ON) in a Chinese cohort.

DETAILED DESCRIPTION:
Patients were sub-divided into an AQP4 seropositive group and an AQP4 seronegative group, according to the results of the AQP4-Ab test. All patients with complete medical histories underwent routine neurological examinations, brain MRIs, and ophthalmological examinations, including best corrected visual acuity (BCVA), intraocular pressure, slit lamp and fundus examination, VF and VEP, laboratory testing, including blood routine, HIV HBV HCV Syphilis, mitochondrial DNA sequencing, and a profile of autoantibodies, including antinuclear antibody (ANA), extractable nuclear antigen antibodies (SSA/SSB), rheumatoid factor (RF), anticardiolipin antibodies (ACA), and antithyroglobulin antibody.

ELIGIBILITY:
Inclusion Criteria:

* Optic neuritis patients

Exclusion Criteria:

* The presence of significant refractive errors (3D of spherical equivalent refraction or 2D of astigmatism), intraocular pressure of 21 mmHg or higher, systemic conditions that could affect the visual system, and a history of ocular trauma or concomitant ocular diseases, including a history of media opacification, ocular pathologies affecting the cornea, lens, retinal disease, glaucoma, or laser therapy. All patients in the study groups had an episode of ON more than six months before the study inclusion time point.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
retinal nerve fiber layer thickness | 2013.11-2016.12

SECONDARY OUTCOMES:
visual field | 2013.11-2016.12
visual evoked potential | 2013.11-2016.12

CONTACTS AND LOCATIONS:
Overall Officials: Hui Yang, Study Director — World Health Organization
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided